CLINICAL TRIAL: NCT04823130
Title: A Multi-center, Exploratory Study to Assess Dupilumab Effect on Pruritus Neuro-mechanisms in Patients With Atopic Dermatitis
Brief Title: Dupilumab Effect on Pruritus Neuro-mechanisms in Patients With Atopic Dermatitis
Acronym: DIFFEREN-STAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LPS16763; 2020-003542-36 (EudraCT Number); U1111-1251-5658 (Other: UTN)
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Results first posted 2023-07-11 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Dermatitis Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: Healthy participants served as control group providing normal skin reference for baseline skin biopsy derived outcome measure and were matched for gender, age, race and anatomical site of skin biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Healthy Participants: Control (No Intervention): Healthy participants with site, age, gender, race, location of targeted lesional and non-lesional skin area matched to selected AD participants, received no treatment, and were considered as a control group.
- Participants With AD: Dupilumab (Experimental): Participants with moderate to severe AD received dupilumab 600 milligrams (mg) subcutaneous (SC) injection on Day 1, followed by dupilumab 300 mg SC injection every 2 weeks (Q2W) from Week 3 to Week 15.
  Interventions: Drug: Dupilumab (SAR231893)

INTERVENTIONS:
Drug: Dupilumab (SAR231893) — Pharmaceutical form: solution for injection Route of administration: subcutaneous
  Other Names: REGN668
  Arms: Participants With AD: Dupilumab

SUMMARY:
Primary Objective:

- Assess change in neuronal architecture following long term treatment with dupilumab in skin biopsies from atopic dermatitis (AD) participants with chronic pruritus.

Secondary Objectives:

* Assess change in neuronal architecture following short term treatment with dupilumab and during follow-up in skin biopsies from AD participants with chronic pruritus.
* To evaluate the efficacy of dupilumab in AD participants with chronic pruritus.
* To evaluate the safety of dupilumab in adult participants with moderate-to-severe AD.

DETAILED DESCRIPTION:
AD participants: A 20-week Observation Period including 16 weeks of treatment for AD participants and a 4-week follow-up period; Healthy participants: 8 days observation period.

ELIGIBILITY:
Inclusion criteria:

For AD participants

* Male or female of greater than or equal to (>=)18 years of age inclusive, at the time of signing the informed consent form (ICF).
* Diagnosed with moderate-to-severe chronic AD for at least 1 year before screening.
* Eligible to be treated with dupilumab according to product monograph.
* Pruritus lasting 6 or more weeks before baseline (Day 1).
* Eczema Area and Severity Index (EASI) score >=12 at baseline.
* Pruritus numerical rating scale (NRS) >=4 at baseline.
* Investigator global assessment (IGA) score of >=3 at screening (on the 0 to 4 scale) at baseline.
* Atopic dermatitis active lesions on the upper limbs or lower limbs suitable for a skin biopsy without oozing, bleeding, or infection on upper limbs or trunk.
* Participants with acute AD lesions as determined by Investigator's judgment.
* Stable treatment with non-prohibited medication or therapy during the study.

For Healthy participants

* Male or female of >=18 years of age inclusive, at the time of signing the ICF.
* Certified as generally healthy by a comprehensive clinical assessment.

Exclusion criteria:

For AD participants

* Previous treatment with dupilumab stopped within 6 months of baseline due to inadequate response to dupilumab.
* Skin conditions other than AD that can confound assessments in the opinion of the investigator.
* Regular use (>2 visits per week) of a tanning booth/parlor within 4 weeks of the Screening Visit.
* Severe concomitant illness(es) that, in the Investigator's judgment, would adversely affect the participant's participation in the study.
* Participants with active tuberculosis (TB) or non-TB mycobacterial infection, or a history of incompletely treated TB unless it is well documented the participant has been adequately treated and can now start treatment with a biologic agent
* Diagnosed with, suspected of, or at high risk of endoparasitic infection, and/or use of antiparasitic drug within 2 weeks before the Screening Visit (Visit 1) or during the Screening Period.
* Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, or antifungals within 2 weeks before the Screening Visit (Visit 1) or during the Screening Period.
* Known or suspected immunodeficiency, including history of invasive opportunistic infections.
* Active malignancy or history of malignancy within 5 years before the Baseline Visit, except completely treated in situ carcinoma of the cervix and completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin.
* Ocular disorder that in the opinion of the Investigator could adversely affect the individual's risk for study participation. Examples include, but are not limited to, individuals with a history of active cases of herpes keratitis, Sjogren's syndrome, keratoconjunctivitis sicca or dry eye syndrome that require daily use of supplemental lubrication or individuals with ocular conditions that require the use of ocular corticosteroids or cyclosporine.
* History of systemic hypersensitivity or anaphylaxis to dupilumab or any other biologic therapy, including any excipient.
* Participant with any other medical or psychological condition including relevant laboratory or electrocardiogram abnormalities at screening.

For healthy participants

* Regular use (>2 visits per week) of a tanning booth/ parlor within 4 weeks of the Screening Visit.
* Treatment with the following concomitant medications and procedures is prohibited within 4 weeks before the Screening Visit or 5 half-lives (whichever is longer) until End of Study Visit:

  * Topical medication
  * Analgesics
  * Immunomodulators
  * Antidepressants
  * Anti-anxiety drugs
* Any Type 2 immune disorders uncontrolled Type 2 diabetes mellitus, Type 1 diabetes mellitus, neuropathy or any other neurological disease.
* Any concomitant illness(es) or conditions that, in the Investigator's judgment, would adversely affect the participant's participation in the study or potentially affect any skin biopsy related read out.
* Positive test for immunoglobulin E (IgE) antibodies.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- United States (2):
  - Investigational Site Number 8400001, Miami, Florida
  - Investigational Site Number 8400002, East Windsor, New Jersey
- Investigational Site Number 2760001, Münster, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS16763 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25290&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 3 active sites in the United States and Germany. A total of 54 participants were enrolled between 22 April 2021 to 30 March 2022.
Pre-assignment Details: Healthy participants were considered as a reference comparator group and received no treatment. Healthy participants underwent only an additional 7-days observational period following collection of the skin biopsy on Day 1 (i.e., up to Day 8). Only safety data was collected for the healthy participants and no other outcome measures were assessed.
Groups:
- Healthy Participants: Control: Healthy participants with site, age, gender, race, location of targeted lesional and non-lesional skin area matched to selected atopic dermatitis (AD) participants, received no treatment, and were considered as a control group.
Period: Overall Study
Arm/Group | Healthy Participants: Control | Participants With AD: Dupilumab
Started | 19 | 35
Safety Population (Safety population included all participants, who actually received at least 1 dose of investigational medicinal product (IMP) or had at least 1 skin biopsy and all healthy participants who had a skin biopsy or another safety assessment performed.) | 13 | 31
Completed | 10 | 28
Not Completed | 9 | 7
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Failure to meet inclusion criteria | 6 | 4
Not completed — Other-unspecified | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on enrolled population.
Groups:
- Participants With AD: Dupilumab: Participants with moderate to severe AD received dupilumab 600 mg SC injection on Day 1, followed by dupilumab 300 mg SC injection Q2W from Week 3 to Week 15.
- Total: Total of all reporting groups
Arm/Group | Healthy Participants: Control | Participants With AD: Dupilumab | Total
Number analyzed (Participants) | 19 | 35 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (14.1) | 41.2 (18.1) | 41.2 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 19 | 32
  Male | 6 | 16 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 33 | 52
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intraepidermal Nerve Fiber Density on Lesional Skin at Week 17
Description: Skin biopsies were used to analyze the epidermal nerve fiber density. Nerve fibers were visualized by staining consecutive sections for the pan-axonal marker protein gene product 9.5 (PGP9.5); and the basement membrane was visualized by staining for collagen type 4. Quantification of intraepidermal nerve fiber density was calculated by assessing nerve fibers crossing the basement membrane per square millimeter (F/mm^2). Data for this outcome measure was not planned to be collected and analyzed for "healthy participant" arm as pre-specified in protocol.
Time Frame: Baseline, Week 17
Population: Analyzed on modified intent-to-treat (mITT) population which included all AD participants who received at least 1 dose of IMP who had at least 1 skin biopsy performed, irrespective of compliance with study protocol and procedures, and who did not use prohibited therapies for AD from screening to end of study. 'Overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: F/mm^2
Arm/Group | Participants With AD: Dupilumab
Number analyzed (Participants) | 27
F/mm^2
  Baseline | 8.4567 (7.2502)
  Change at Week 17: number analyzed (Participants) | 20
  Change at Week 17 | 4.2618 (6.7538)

2. Primary Outcome: Percentage of Participants With Change From Baseline in Nerve Fiber Branching on Lesional Skin at Week 17
Description: Skin biopsies were used to analyze the epidermal nerve fiber branching. Nerve fibers were visualized by staining consecutive sections for the pan-axonal marker PGP9.5; and the basement membrane was visualized by staining for collagen type 4. Branching of epidermal nerve fibers was assessed semi-quantitatively by classifying participants into 4 groups depending on the predominant intraepidermal nerve fiber branching pattern as follows: only linear (100% linear), mainly linear (>60% linear), mainly branched (>60% branched), only branched (100% branched). Percentage of participants with change in nerve fiber branching status from baseline on lesional skin at Week 17 are reported in this outcome measure.
Time Frame: Baseline, Week 17
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for "healthy participant" arm as pre-specified in protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With AD: Dupilumab
Number analyzed (Participants) | 15
percentage of participants
  Only linear | 0
  Mainly linear | 60.0
  Mainly branched | 40.0
  Only branched | 0

3. Secondary Outcome: Change From Baseline in Intraepidermal Nerve Fiber Density on Lesional Skin at Weeks 3 and 21
Description: Skin biopsies were used to analyze the epidermal nerve fiber density. Nerve fibers were visualized by staining consecutive sections for the pan-axonal marker PGP9.5; and the basement membrane was visualized by staining for collagen type 4. Quantification of intraepidermal nerve fiber density was calculated by assessing nerve fibers crossing the basement membrane per square millimeter (F/mm^2).
Time Frame: Baseline, Weeks 3 and 21
Population: Data was not collected and analyzed for this outcome measure as no optional skin biopsies were done at Weeks 3 and 21.
Arm/Group | Participants With AD: Dupilumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline in Nerve Fiber Branching on Lesional Skin at Weeks 3 and 21
Description: Skin biopsies were used to analyze the epidermal nerve fiber branching. Nerve fibers were visualized by staining consecutive sections for the pan-axonal marker PGP9.5; and the basement membrane was visualized by staining for collagen type 4. Branching of epidermal nerve fibers was assessed semi-quantitatively by classifying participants into 4 groups depending on the predominant intraepidermal nerve fiber branching pattern as follows: only linear (100% linear), mainly linear (>60% linear), mainly branched (>60% branched), only branched (100% branched).
Time Frame: Baseline, Weeks 3 and 21
Population: Data was not collected and analyzed for this outcome measure as no optional skin biopsies were done at Weeks 3 and 21.
Arm/Group | Participants With AD: Dupilumab
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in Peak Pruritus Assessed by Numeric Rating Scale (NRS) Scores at Weeks 17 and 21
Description: Peak Pruritus NRS was an assessment tool used to report the intensity of participant's pruritus (itch) during a daily recall period. Participants were asked to rate their worst itch on a 0 ("No itch") to 10 ("Worst itch imaginable") NRS by answering the following question: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". Higher scores indicated greater severity.
Time Frame: Baseline, Weeks 17 and 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With AD: Dupilumab
Number analyzed (Participants) | 7
score on a scale
  Week 17 | -6.6 (3.6)
  Week 21 | -7.4 (1.4)

6. Secondary Outcome: Change From Baseline in Eczema and Severity Index (EASI) Total Score at Weeks 17 and 21
Description: EASI was a validated measure used to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, and edema], scratching [excoriation], and lichenification) were each assessed for severity by the Investigator on a scale of "0" (absent) through "3" (severe). EASI area score was based upon percent (%) body surface area (BSA) with AD in each body region: 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), and 6 (90% to 100%). Total EASI score was derived as the sum of the 4 region scores and ranged from 0 (minimum) to 72 (maximum). Higher scores indicated greater severity of AD.
Time Frame: Baseline, Weeks 17 and 21
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for "healthy participant" arm as pre-specified in protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With AD: Dupilumab
Number analyzed (Participants) | 12
score on a scale
  Week 17 | -18.9 (6.4)
  Week 21: number analyzed (Participants) | 10
  Week 21 | -19.5 (6.4)

7. Secondary Outcome: Change From Baseline in Scoring Atopic Dermatitis (SCORAD) Total Score at Weeks 17 and 21
Description: SCORAD was used to standardize the extent and severity of AD. It consisted of 3 components i.e., A =extent or affected BSA assessed as a % of each defined body area and reported as sum of all areas, with a maximum score of 100%. B=severity of 6 specific symptoms of AD (redness, swelling, oozing/crusting, excoriation, skin thickening/lichenification, dryness) assessed using following scale: none (0), mild (1), moderate (2), or severe (3) (for a maximum of 18 total points) and C=subjective symptoms scored by participants on VAS, where "0"=no itch (or no sleeplessness) and "10"=worst imaginable itch (or sleeplessness) with a maximum score of 20. SCORAD total score was calculated using these 3 aspects: extent (A: 0-100), severity (B: 0-18), and subjective symptoms (C: 0-20) using the formula: A/5 + 7*B/2+ C. SCORAD total score ranged from 0 to 103, where 0 = no disease to 103 = severe disease. Higher values of SCORAD represent worse outcome.
Time Frame: Baseline, Weeks 17 and 21
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With AD: Dupilumab
Number analyzed (Participants) | 19
score on a scale
  Week 17 | -77.2 (32.3)
  Week 21: number analyzed (Participants) | 15
  Week 21 | -81.3 (35.0)

8. Secondary Outcome: Change From Baseline in Patient-Reported Outcomes Measurement Information (PROMIS-itch) Itch-Severity Total Score at Weeks 17 and 21
Description: PROMIS-itch represents a novel suite of participant-reported outcome (PRO) measures for the itch. The PROMIS-Itch severity score consists of 7 questions: 4 questions scored on a scale of 1 to 5: 1) How intense was your itch at its worst; 2) How intense was your itch in general; 3) What is your level of itch right now; 4) How often did you feel the itch; and rest 3 questions (same questions as 1 to 3 mentioned before but scaled on a scale of 0 to 10) were scored on a scale of 0 to 10. Higher scores for each question indicated worse outcome. The total PROMIS-itch score was calculated as the sum of the 7 questions and ranged from 4 (better outcome) to 50 (worse outcome), where a higher score indicated worse condition.
Time Frame: Baseline, Weeks 17 and 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With AD: Dupilumab
Number analyzed (Participants) | 13
score on a scale
  Week 17 | -30.8 (9.0)
  Week 21 | -28.8 (11.5)

9. Secondary Outcome: Change From Baseline in Patient Oriented Eczema Measure (POEM) Total Score at Weeks 17 and 21
Description: The POEM was a 7-item, validated questionnaire used in clinical practice and clinical trials to assess disease symptoms in children and adults with AD. The format is participant response to 7 items (dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping) based on symptom frequency during the past week (i.e., 0 = 'no days', 1 = '1 to 2 days', 2 = '3 to 4 days', 3 = '5 to 6' days, and 4 = 'every day'). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (severe disease). Higher scores indicated more severe disease and poor quality of life.
Time Frame: Baseline, Weeks 17 and 21
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With AD: Dupilumab
Number analyzed (Participants) | 14
score on a scale
  Week 17 | -17.2 (5.3)
  Week 21: number analyzed (Participants) | 13
  Week 21 | -16.1 (5.9)

10. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score at Weeks 17 and 21
Description: DLQI was a 10-item PRO questionnaire that measured the impact of AD disease symptoms and treatment on quality of life. Each question was evaluated on a 4-point scale ranged from 0 to 3 where, 0 = not at all, 1= a little, 2= a lot, 3= very much, where higher scores indicated more impact on quality of life. Scores from all 10 questions were added up to give DLQI total score that ranged from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of participants.
Time Frame: Baseline, Weeks 17 and 21
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With AD: Dupilumab
Number analyzed (Participants) | 17
score on a scale
  Week 17 | -16.1 (7.4)
  Week 21: number analyzed (Participants) | 16
  Week 21 | -14.8 (8.1)

11. Secondary Outcome: Change From Baseline in Atopic Dermatitis Control Tool (ADCT) Total Score at Weeks 17 and 21
Description: ADCT was a PRO questionnaire designed to assess participant-self-perceived control of their eczema. ADCT contained 6 items allowing a comprehensive coverage of the dimensions defining AD control, i.e., overall severity of AD symptoms, frequency of intense episodes of itching, extent of AD related bother, impact on sleep, impact on daily activities, impact on mood or emotions. Each item of the ADCT is rated from 0 (no problem) to 4 (worst) Likert scale and is equally weighted. The sum of the 6 items gives the total score that ranged from 0 (best disease control) to 24 (worst disease control). Higher scores indicate lower AD control.
Time Frame: Baseline, Weeks 17 and 21
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With AD: Dupilumab
Number analyzed (Participants) | 14
score on a scale
  Week 17 | -17.9 (4.1)
  Week 21 | -15.9 (6.2)

12. Secondary Outcome: Change From Baseline in Sleep Quality Numerical Rating Scale Score at Weeks 17 and 21
Description: Sleep quality NRS was used to assess the quality of the participant's previous night's sleep using a 0 ("Worst possible sleep") to 10 ("Best possible sleep") NRS. Participants were asked to complete the following question upon awakening: "Select the number (0 to 10) that best describes the quality of your sleep last night". Higher score indicated better outcome.
Time Frame: Baseline, Weeks 17 and 21
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With AD: Dupilumab
Number analyzed (Participants) | 5
score on a scale
  Week 17: number analyzed (Participants) | 3
  Week 17 | 0.7 (5.0)
  Week 21 | 3.0 (5.4)

13. Secondary Outcome: Change From Baseline in Skin Pain Numerical Rating Scale Score at Weeks 17 and 21
Description: Skin pain NRS was used to assess participant's skin pain at its worst in the past 24 hours using a 0 ("Not at all") to 10 ("Very much") NRS. Participants were asked the following question: "Think about all the areas of your skin with eczema. How much did your skin burn at its worst in the past 24 hours?" Lower score indicated better outcome.
Time Frame: Baseline, Weeks 17 and 21
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With AD: Dupilumab
Number analyzed (Participants) | 4
score on a scale
  Week 17: number analyzed (Participants) | 3
  Week 17 | -5.3 (2.9)
  Week 21 | -5.3 (2.2)

14. Secondary Outcome: Change From Baseline in Skin Sensitivity Numerical Rating Scale Score at Weeks 17 and 21
Description: Skin sensitivity NRS was a 1 item PRO measure asking the participants to rate their skin sensitivity to touch using a 0 ("Normal") to 10 ("Extremely sensitive") NRS. Participants were asked the following question: "Think about all the areas of your skin with eczema. How sensitive was your skin at its worst in the past 24 hours?" Lower score indicated better outcome.
Time Frame: Baseline, Weeks 17 and 21
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With AD: Dupilumab
Number analyzed (Participants) | 4
score on a scale
  Week 17: number analyzed (Participants) | 3
  Week 17 | -7.7 (1.5)
  Week 21 | -7.3 (2.2)

15. Secondary Outcome: Change From Baseline in Skin Burning Numerical Rating Scale Score at Weeks 17 and 21
Description: Skin burning NRS was a 1-item PRO measure asking participants to rate the burning sensation of their skin in the past 24 hours using a 0 ("Not at all") to 10 ("Very much") NRS. Participants were asked the following question: "Think about all the areas of your skin with eczema. How much did your skin burn at its worst in the past 24 hours?" Lower score indicated better outcome.
Time Frame: Baseline, Weeks 17 and 21
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With AD: Dupilumab
Number analyzed (Participants) | 4
score on a scale
  Week 17: number analyzed (Participants) | 3
  Week 17 | -4.3 (1.5)
  Week 21 | -5.5 (2.9)

16. Secondary Outcome: Percentage of Participants With Change of Greater Than or Equal to (>=4) Point in Pruritus Numerical Rating Scale From Baseline at Weeks 17 and 21
Description: Pruritus NRS was an assessment tool used to report the intensity of participant's pruritus (itch) during a daily recall period. Participants were asked to rate their worst itch on a 0 ("No itch") to 10 ("Worst itch imaginable") NRS by answering the following question: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?". Higher scores indicated greater severity. Percentage of participants with change of >=4 point in pruritus NRS scale from baseline at Weeks 17 and 21 are reported in this outcome measure.
Time Frame: Baseline, Weeks 17 and 21
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Participants With AD: Dupilumab
Number analyzed (Participants) | 7
percentage of participants
  Week 17 | 0
  Week 21 | 0

ADVERSE EVENTS:
Time Frame: For Dupilumab group participants: from first dose (i.e., Day 1) of IMP administration up to end of study visit (i.e., up to Week 21). For healthy participants: from Baseline up to end of study for healthy participants group (i.e., at Day 8)
Description: Analysis was performed on safety population.
Arm/Group | Healthy Participants: Control | Participants With AD: Dupilumab
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/31
Other Adverse Events (participants affected / at risk) | 0/13 | 24/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Participants: Control (N=13) | Participants With AD: Dupilumab (N=31)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Participants: Control (N=13) | Participants With AD: Dupilumab (N=31)
Asymptomatic Covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 2 (2)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Oral Herpes (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Suspected Covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Tinea Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 7 (9)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (2)
Conjunctivitis Allergic (Eye disorders) | 0 (0) | 1 (1)
Eye Pruritus (Eye disorders) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain Of Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Injection Site Mass (General disorders) | 0 (0) | 1 (1)
Injection Site Swelling (General disorders) | 0 (0) | 1 (1)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT04823130/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT04823130/SAP_001.pdf